CLINICAL TRIAL: NCT04633720
Title: Exploration of the Appropriate Combination of Positive End Expiratory Pressure and Tidal Volume Using the Intratidal Compliance-volume Profile in Children
Brief Title: Exploration of the Appropriate Combination of Positive End Expiratory Pressure and Tidal Volume Using the Intratidal Compliance Volume Profile in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H2009-175-1162
Record Dates: First submitted 2020-11-08; First posted 2020-11-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Compliance
MeSH Terms: interventions — Positive-Pressure Respiration; Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of intratidal compliance (Experimental): When the patient is in the supine position 10 minutes after induction of anesthesia, the following 4 mechanical ventilator settings are applied to the patients in order.
  1. Positive end-expiratory pressure 8 cmH2O, tidal volume 8 ml/kg
  2. Positive end-expiratory pressure 10 cmH2O, tidal volume 5 ml/kg
  3. Positive end-expiratory pressure 10 cmH2O, tidal volume 8 ml/kg
  4. Positive end-expiratory pressure 12 cmH2O, tidal volume 5 ml/kg
  Interventions: Other: Changes in positive end-expiratory pressure and tidal volume

INTERVENTIONS:
Other: Changes in positive end-expiratory pressure and tidal volume — When the patient is in the supine position 10 minutes after induction of anesthesia, the following 4 mechanical ventilator settings are applied to the patients in order.
  Positive end-expiratory pressure 8 cmH2O, tidal volume 8 ml/kg Positive end-expiratory pressure 10 cmH2O, tidal volume 5 ml/kg Positive end-expiratory pressure 10 cmH2O, tidal volume 8 ml/kg Positive end-expiratory pressure 12 cmH2O, tidal volume 5 ml/kg

SUMMARY:
In children under 6 years of age undergoing regular surgery during general anesthesia, the intratidal compliance profile is evaluated when different tidal volumes are applied at different positive end expiratory pressures.

Then determine the most appropriate combination of positive end-tidal pressure and tidal volume.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing surgery > 1 hour under general anesthesia
* Children ≤ 6 years
* American society of anesthesiology physical status I, II

Exclusion Criteria:

* Previous lung surgery
* Bronchopulmonary dysplasia, respiratory distress syndrome
* Other interstitial lung disease
* Laparoscopic surgery
* Thoracic surgery, abdominal surgery

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Intratidal compliance profiles in each ventilator settings | During general anesthesia (up to about 50 min-1 hr after induction of anesthesia)
  The investigators will determine Intratidal compliance profile using the changes in compliance over time
  --> I, merely increasing compliance profile; IH, increasing turning into horizontal compliance profile; D, merely decreasing compliance profile; HD, horizontal turning into decreasing compliance profile; IHD, increasing turning into horizontal and further turning into decreasing compliance profile If compliance profile is I, the PEEP is low. On the other hand, compliance profile is D, PEEP level is considered to be high.

SECONDARY OUTCOMES:
Respiratory compliance | During general anesthesia (up to about 50 min-1 hr after induction of anesthesia)
  ml cmH2O-1
Driving pressure | During general anesthesia (up to about 50 min-1 hr after induction of anesthesia)
  cmH2O
Blood pressure | During general anesthesia (up to about 50 min-1 hr after induction of anesthesia)
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Kang P, Song IS, Ji SH, Lee HC, Jang YE, Kim EH, Kim HS, Kim JT. Determining optimal positive end-expiratory pressure and tidal volume in children by intratidal compliance: a prospective observational study. Br J Anaesth. 2022 Jan;128(1):214-221. doi: 10.1016/j.bja.2021.09.024. Epub 2021 Oct 20. PMID 34686309